CLINICAL TRIAL: NCT00105222
Title: Evaluation of Systemic Nitrite Infusion and Its Effect on Exercise Physiology and Metabolism
Brief Title: Effect of Nitrite on Exercise Physiology and Metabolism
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050114; 05-H-0114
Record Dates: First submitted 2005-03-09; First posted 2005-03-10 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2013-08-16

CONDITIONS: Healthy; Healthy Volunteer; HV
Keywords: Cycle Ergometer; Exercise Physiology; Nitric Oxide; Sodium Nitrite; Healthy Volunteers; Normal Volunteer; Healthy Volunteer; HV
MeSH Terms: interventions — Sodium Nitrite

INTERVENTIONS:
Drug: Sodium Nitrite

SUMMARY:
This study will examine how nitrite infusions affect exercise tolerance (how much a person can exercise before having to stop). Exercise ability is limited by how fast oxygen can be delivered to the body and how fast the body can produce energy. Both of these processes are affected by nitric oxide (NO), a gas produced by cells that line blood vessels. NO is important in regulating blood vessel dilation, and consequently, blood flow. Nitrite may act as a storehouse for nitric oxide and be able to improve exercise tolerance.

Healthy normal volunteers between 21 and 45 years of age who can use an exercise bicycle may be eligible for this study. Candidates are screened with a medical history, physical examination, electrocardiogram, breathing tests, blood tests, and a pregnancy test for women who are able to bear children. Pregnant women are excluded from the study. The screening session includes practice exercise on the bicycle.

Participants exercise on a stationery exercise bicycle for about 30 minutes on each of two study days. During the test, they breathe in and out of a mouthpiece that allows inhaled and exhaled respiratory gases to be measured. Before subjects begin to exercise, a small tube is placed in the artery of their forearm inside the elbow. A longer tube called a central line is placed in a deeper vein in the neck after the area has been numbed. A thinner tube, called a pulmonary artery catheter, is placed through the central line and advanced into the chambers of the heart, through the heart valve, and into the lung artery. This catheter measures various pressures directly in the heart and lungs. Blood samples are drawn through the catheter also, to avoid the need for multiple needle sticks. Another tube is placed in the vein of the other arm to deliver medications.

Thirty minutes after all the tubes are placed, a blood sample is drawn for baseline measurements. Then, either saline (sterile salt water) or nitrite is injected into the tube in the arm vein. Thirty minutes after the injection, the subject starts exercising on the bicycle. The work setting on the bicycle is increased every minute, and the subject pedals until he or she is too tired to continue. During the test, a small blood sample is collected every 2 minutes. Heart rate, blood pressure, and heart rhythms are continuously monitored.

After the test on the first day, participants are admitted to the hospital to rest for the remainder of the afternoon and evening. The tubes are kept in place for the following morning, when the procedure is repeated exactly as before, except that subjects who received saline the first day are given nitrite the second day, and vice versa.

...

DETAILED DESCRIPTION:
During exercise, there is a lag in the rate at which oxygen uptake (VO2) rises to meet energy demand. It is uncertain whether this limitation is due to inadequate O2 delivery to working muscle, limitations to the rate at which mitochondria can generate ATP to meet demand, or by a combination of both. Both of these limitations may be modulated by nitric oxide. Nitric oxide (NO) has been implicated in numerous physiological functions, including control of skeletal muscle vasodilation and oxidative metabolism. During exercise, NO will both vasodilate skeletal muscle and modulate (inhibit) mitochondrial respiration. The latter effect could either decrease oxygen extraction by limiting the ability of mitochondria to utilize oxygen, or paradoxically increase oxygen utilization by inhibiting mitochondria proximal to blood vessels, an effect that facilitates oxygen diffusion to distal tissue and mitochondria (NO dependent facilitated oxygen diffusion). Previous studies have demonstrated that NO production increases during exercise and regional inhibition of NO production from endothelial NO synthase reduces exercise-dependent blood flow by approximately 10%. NOS inhibitors such as N(G) -nitro-L-arginine methyl ester (L-NAME) have been shown to decrease exercise tolerance, and NO precursors (L-arginine) to increase exercise tolerance. Administration of inhaled NO during exercise has not been shown to increase exercise tolerance.

Considering the potential role of nitrite bioconversion to NO during hypoxia, is likely that nitrite plays an important role in modulating exercise physiology. We therefore hypothesize that during aerobic, and in particular anaerobic exercise, erythrocyte and plasma nitrite will be converted to NO and modulate muscle blood flow, mitochondrial respiration, oxygen diffusion and ultimately maximal oxygen consumption. While we expect these effects will increase maximal oxygen consumption and increase work output, it is also distinctly possible that NO production from nitrite during exercise will inhibit mitochondrial respiration and decrease maximal oxygen consumption. The purpose of the present study is to investigate the effects of aerobic-to-anaerobic exercise on circulating nitrite stores in erythrocytes and plasma in the arterial and central venous circulation and the effects of systemic nitrite infusion on aerobic and anaerobic exercise capacity. Physiological parameters including maximal oxygen consumption (VO2max), maximal CO2 and NO production (VCO2max and VNOmax), maximal work, rate of perceived exertion (RPE), anaerobic threshold, and pulmonary gas exchange (VO2, VCO2, VE) will be monitored during exercise with and without nitrite infusions. Our primary endpoint will be VO2 max with nitrite infusion compared to VO2 max with saline placebo infusion.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects must be 21-45 years of age.

Subject must be in good health and able to perform cycle ergometry for the length of the study.

Subjects must provide informed, written consent for participation in this study.

Female subjects of childbearing age must have a negative pregnancy test.

EXCLUSION CRITERIA:

Subjects with a history of cardiac, pulmonary, peripheral vascular, or mitochondrial disease.

Subjects with abnormal EKG other than sinus bradycardia.

Individuals with a future cardiovascular risk greater than 1 % in the next 10 years will be excluded from the study. Risk will be calculated using the Framingham risk calculator published on the web site: http://hin.nhlbi.nih.gov/atpiii/calculator.asp?usertype=prof.

Subjects with any physical condition (for example, knee problems) that may impair their performance during exercise testing.

Subjects who have a history of smoking within one year.

Subjects with anemia (defined as hemoglobin less than 10 g/dL).

Subjects with a history of reaction to a medication or other substance characterized by dyspnea and cyanosis will not participate in this study.

Subjects with G6PD deficiency.

Subjects with a baseline methemoglobin level greater than 1%.

Lactating females who are breastfeeding, will not participate since nitrite crosses into breast milk and could cause methemoglobinemia in the infant.

No volunteer subject will be allowed to take any medication (oral contraceptive agents are allowed), vitamin supplements, herbal preparations, nutriceuticals or other alternative therapies for at least one month prior to study and will not be allowed to take aspirin or NSAIDs for one week prior to study.

Subjects with a blood pressure of less than 100/70 mmHg on the study day will be excluded from the protocol.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2005-03-08; Primary Completion 2013-08-16 (Actual); Study Completion 2013-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Kato, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Beckman JS, Koppenol WH. Nitric oxide, superoxide, and peroxynitrite: the good, the bad, and ugly. Am J Physiol. 1996 Nov;271(5 Pt 1):C1424-37. doi: 10.1152/ajpcell.1996.271.5.C1424. PMID 8944624
- [Background] Boucher JL, Moali C, Tenu JP. Nitric oxide biosynthesis, nitric oxide synthase inhibitors and arginase competition for L-arginine utilization. Cell Mol Life Sci. 1999 Jul;55(8-9):1015-28. doi: 10.1007/s000180050352. PMID 10484661
- [Background] Furchgott RF, Zawadzki JV. The obligatory role of endothelial cells in the relaxation of arterial smooth muscle by acetylcholine. Nature. 1980 Nov 27;288(5789):373-6. doi: 10.1038/288373a0. PMID 6253831